CLINICAL TRIAL: NCT01183806
Title: Effects of Exercise and Rivastigmine on Quality of Life of Alzheimer's Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Ailton de Souza Melo, Ailton de Souza Melo,PhD, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PA-01
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Exercise; Rivastigmine; Quality of life
MeSH Terms: conditions — Alzheimer Disease; Motor Activity | interventions — Rivastigmine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rivastigmine and exercise program (Experimental): Experimental group: Rivastigmine and exercise program: All patients will monthly receive Rivastigmine (Exelon patch). The exercise training program consists of two 40-minute sessions per week for six months and includes aerobic, strength, flexibility and balance training
  Interventions: Drug: Rivastigmine; Other: Exercise training program
- Rivastigmine (Active Comparator): Control group : Rivastigmine All patients will monthly receive Rivastigmine (Exelon patch)
  Interventions: Drug: Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine — All patients start on a 5-cm2 rivastigmine transdermal patch and their dose is progressively increased
  Other Names: Rivastigmine use
Other: Exercise training program — Exercise training program
  Other Names: Rivastigmine use and exercise program
  Arms: Rivastigmine and exercise program

SUMMARY:
The purpose of this study is to determine whether a exercise program when combined with rivastigmine (Exelon patch) drug treatment compared with rivastigmine drug treatment alone would improve quality of life, ability to perform activities of daily living (ADL) and cognition in patients with Alzheimer's disease.

Hypothesis:

Ho: Rivastigmine drug treatment combined with exercise is not superior to rivastigmine drug treatment to improve quality of life of Alzheimer's disease patients.

H1: Rivastigmine drug treatment combined with exercise is superior to rivastigmine drug treatment to improve quality of life of Alzheimer's disease patients, with an expectative of 15% of improvement in the quality of life scale measurement

DETAILED DESCRIPTION:
After screening and informed consent, that will be collected demographical data from patient. Another researcher will evaluate the cognition, through MMSE; the activities of daily living, through Activities of Daily Living Questionnaire of Alzheimer disease; patient and caregiver's quality of life through Quality of life scale in Alzheimer's disease (QOL-AD); functional mobility, through Time Up and Go test.

Afterwards, the pharmacist will give the medicine, orientations about its administration and clarify possible doubts. Therapy will begin with the small patch of 5 mg/24 h and, if well tolerated, the dose will be increased to the 10 mg/24 h patch.

The patients will be randomly assigned, through a computer program list, to exercise or control group. The patient and caregiver exercise group will receive information about the two-day/week exercise program at physiotherapy ambulatory. Monthly, all patients and caregiver will be clinically reevaluated during six months.

The forty minutes exercise program will include aerobic, strength, flexibility and balance training, organize in the follow sequence:

- Ten minutes of global stretching (shoulder girdle, upper limbs, lower limbs and trunk) along the beginning and final of the session. Each stretch posture will last 30 seconds.

Alternation of A and B sessions, lasting 30 minutes:

* Session A: Aerobic training on treadmill. Progression of 10 to 30 minutes of continuous aerobic activity
* Session B: - Resisted kinesiotherapy (strength training) with use of weights to be attached around the ankles and wrist of initially 1 Ib. The physiotherapist will evaluate if patient can progress to a higher weight during sessions.
* Walking over obstacles on the ground and direction change with use of cones.
* Functional activities like transfer exercise (stand/sit exercise) and squatting The monitoring of the exercise, its progress and any other observation will be register in a control form by the physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of probable Alzheimer's disease
* At least 55 years of age
* Same caregiver (familiar or paid one) for at least 3 months before, who is able to follow the patient in a two-day/week exercise program
* Do not be taking other prescribed medication for Alzheimer disease
* Treated stable hypertension

Exclusion Criteria:

* Mini-Mental State Examination (MMSE) score of less than 12
* Can't follow simple commands;
* Can't answer two or more items of Quality of life questionnaire
* Practiced regular exercise or physiotherapy/ occupational therapy in the last two months.
* Diagnosed psychiatric condition (including depression).
* Use of neuroleptic drugs
* Orthopedic, neurologic, or behavioral limitations that may preclude exercise training
* Visual or hearing impairment that may preclude exercise training or comprehension

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Patients' Quality of life | Monthly for six months
  Patients' Quality of life of assessed by Quality of life scale in Alzheimer's disease (QOL-AD)- Portuguese version

SECONDARY OUTCOMES:
Cognition | Monthly for six months
  Cognition change, through Mini-Mental State examination (MMSE)
Caregivers' Quality of life | Monthly for six months
  Caregivers' Quality of life of assessed by Quality of life scale in Alzheimer's disease (QOL-AD)- Portuguese version
Activities of daily living | Monthly for six months
  Activities of daily living, through Activities of Daily Living Questionnaire of Alzheimer disease - portuguese version
Functional mobility | Monthly for six months
  Functional mobility, through Time Up and Go test

CONTACTS AND LOCATIONS:
Overall Officials: Paula Aguiar, Study Chair — Federal University of Bahia
Locations (2):
- Brazil (2):
  - Ferderal University of Bahia - DINEP, Salvador, Estado de Bahia
  - Federal University of Bahia, Salvador, Estado de Bahia

REFERENCES:
- [Derived] Aguiar P, Monteiro L, Feres A, Gomes I, Melo A. Rivastigmine transdermal patch and physical exercises for Alzheimer's disease: a randomized clinical trial. Curr Alzheimer Res. 2014;11(6):532-7. doi: 10.2174/1567205011666140618102224. PMID 24938502